CLINICAL TRIAL: NCT00025207
Title: A Phase II Study Of ZD 1839 (NSC 715055, IND 61187) In Patients With Malignant Mesothelioma
Brief Title: Gefitinib in Treating Patients With Malignant Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02414; CLB-30101; U10CA031946 (NIH); CDR0000068938 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-10-11; First posted 2003-09-10 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Advanced Malignant Mesothelioma; Epithelial Mesothelioma; Recurrent Malignant Mesothelioma; Sarcomatous Mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant; Solitary Fibrous Tumor, Pleural | interventions — Gefitinib

ARMS (1):
- Treatment (gefitinib) (Experimental): Patients receive oral gefitinib once daily on days 1-21. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gefitinib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: gefitinib — Given orally
  Other Names: Iressa; ZD 1839
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of gefitinib in treating patients who have malignant mesothelioma. Biological therapies such as gefitinib may interfere with the growth of the tumor cells and slow the growth of malignant mesothelioma

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the activity of gefitinib, in terms of failure-free survival, in patients with malignant mesothelioma.

II. Determine the response rate in patients treated with this drug. III. Determine the toxicity of this drug in these patients. IV. Determine the overall survival of patients treated with this drug. V. Determine whether overexpression of epidermal growth factor receptor and expression of cyclo-oxygenase-2 can predict the effectiveness of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral gefitinib once daily on days 1-21. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months for 1 year and then every 6 months for up to 3 years.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 7-10 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignant mesothelioma that is not amenable to curative surgery or radiotherapy

  * Epithelial, sarcomatoid, or mixed subtype
  * Any site of origin (including, but not limited to, the pleura, peritoneum, pericardium, or tunica vaginalis) allowed
* Measurable disease, defined as lesions that can be accurately measured in at least 1 dimension (longest diameter) as at least 20 mm with conventional techniques or at least 10 mm with spiral CT scan

  * Must be outside prior radiation port
  * Lesions not considered measurable include the following:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Abdominal masses not confirmed and followed by imaging techniques
    * Cystic lesions
* No known brain metastases
* Performance status - CTC 0-1
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT no greater than 2.5 times ULN
* Creatinine no greater than 1.5 times ULN
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other concurrent active malignancy except nonmelanoma skin cancer

  * Disease considered not currently active if completely treated with less than a 30% risk for relapse
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No prior epidermal growth factor receptor-inhibitor therapy
* Prior intrapleural cytotoxic or sclerosing agents (including bleomycin) allowed
* No prior systemic cytotoxic chemotherapy for malignant mesothelioma
* No concurrent chemotherapy
* At least 1 week since prior CYP3A4 inducers (e.g., dexamethasone, glucocorticoids, progesterone)
* No concurrent CYP3A4 inducers (e.g., dexamethasone)
* No concurrent hormonal therapy (e.g., tamoxifen) except steroids for adrenal failure or hormones for non disease-related conditions (e.g., insulin for diabetes)
* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy, including for palliation
* See Disease Characteristics
* At least 2 weeks since prior major surgery
* At least 1 week since other prior CYP3A4 inducers (e.g., carbamazepine, ethosuximide, griseofulvin, nafcillin, nelfinavir mesylate, nevirapine, oxcarbazepine, phenobarbital, phenylbutazone, phenytoin, primidone, rifabutin, rifampin, rofecoxib, St. John's Wort, sulfadimidine, sulfinpyrazone, or troglitazone)
* No other concurrent CYP3A4 inducers
* No concurrent CYP3A4 substrates or inhibitors
* No other concurrent investigational agent
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No concurrent chlorpromazine, amiodarone, or chloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-09; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Percentage of patients who remain failure-free | Time between the initiation of treatment and initial failure (disease progression, relapse, death), assessed up to 3 months
  Kaplan-Meier's product limit estimator and curves will be used.

SECONDARY OUTCOMES:
Tumor response rate | Up to 4 years
  An exact binomial confidence interval will be generated.
Toxicities, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v3.0 | Up to 4 years
  For each type of toxicity experienced, the frequency of reported toxicity will be summarized by the most severe grade.
Overall survival | Up to 4 years
  Kaplan-Meier's product limit estimator and curves will be used.
Failure-free survival within patient subgroups defined in terms of epidermal growth factor receptor (EGFR) overexpression and cyclooxygenase-2 (COX-2) expression | Up to 4 years
  An exact binomial confidence interval will be generated.

CONTACTS AND LOCATIONS:
Overall Officials: Ramaswamy Govindan, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States